CLINICAL TRIAL: NCT01722903
Title: Perioperative Detection and Characterization of Circulating Tumor Cells in Patients Undergoing Colorectal Cancer Liver and Lung Metastasectomy
Brief Title: Detection of CTCs in Patients Undergoing Surgery for Stage IV Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Angela Lehman, HRT3, Milton S. Hershey Medical Center
Other Study IDs: 39748EP
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Stage IV Colorectal Cancer; Liver Metastases; Lung Metastases
Keywords: colorectal cancer; liver metastases; lung metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Colorectal liver and lung metastases, adjacent healthy liver and lung metastases, isolated circulating tumor cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stage IV colorectal cancer: CTCs will be drawn during liver and/or lung metastasectomy for colorectal cancer

SUMMARY:
Colorectal cancer (CRC) is the second leading cause of cancer deaths in the United States. About 90% of CRC related deaths are due to metastatic spread-mostly to the liver and lungs. With adequate multidisciplinary patient selection, CRC liver and lung metastasectomy significantly improves survival and offers the best chance for a cure. However, patients with limited lung or liver metastases are clinically underserved and poorly scientifically studied. The individual indication for resection and the decision making for adjuvant systemic therapies remains a challenge. More sensitive techniques to detect occult disease are needed for metastatic CRC (mCRC) patients, and perioperative analysis of circulating tumor cells (CTCs) may provide an outstanding opportunity to develop such innovative methods. We hypothesize that CTCs are enriched during CRC liver and/or lung metastasectomy, and that they can be isolated and characterized in an attempt to identify novel therapeutic targets.

CTCs are believed to be causing metastasis and may provide a non-invasive alternative to organ biopsies for the detection, characterization and monitoring of solid cancers. CTC numbers have been shown to be a strong predictor of Progression Free Survival and Overall Survival for mCRC patients. The CellSearch system (Veridex LLC, Ratinas, NJ, USA) currently is the only FDA approved test for the evaluation of CTC numbers in metastatic breast, prostate and colorectal cancer. However, the rarity of CTCs in the blood leads to limited capture efficiency and the CellSearch system fixes cells, preventing further molecular characterization of CTCs by functional assays and primary cell culture. In this protocol the CellSearch system will be compared to a new technology, called the Flexible Micro Spring Array (FMSA) device, developed by Dr. Zheng, Department of Bioengineering, Penn State University, University Park. This novel approach enables size-exclusion based filtration for viable CTC enrichment. The FMSA device is inexpensive, works rapidly, and retains viable CTCs for further biological study. Using both the CellSearch system and the FMSA device, we will determine the kinetics of CTC shedding into circulation, develop an effective system for isolation, enumeration, and further enrichment CTCs, and use this system to find characteristics of different CTC populations.

DETAILED DESCRIPTION:
More sensitive techniques to detect occult disease are needed for metastatic CRC (mCRC) patients, and perioperative analysis of circulating tumor cells (CTCs) may provide an outstanding opportunity to develop such innovative methods.

Determine kinetics of CTC shedding into the circulation: Perioperative CTC detection has the potential to explain how and when CTCs are shed into the blood. Findings could explain the nature of CTCs with important impact on understanding metastatic spread and relevant clinical applications.

Since this protocol includes blood draws at multiple time points at different distances from the metastases, results could further clarify if the rarity or absence of CTCs in the peripheral blood of some mCRC patients can be explained by dilution. Comparison of patients with CRC liver to lung metastases might help explain different patterns of organ spread. Results of this study could establish CTCs as a prognostic biomarker identifying candidates who will benefit from metastasectomy or for those who are candidates for additional or palliative systemic treatments because of a high risk for later recurrence.

* Develop effective system for isolation, enumeration, enrichment and further characterization of live CTCs: One of the current issues of CTC analysis is the enrichment of those rare cells from blood. We plan to analyze perioperatively drawn blood using the flexible micro spring array (FMSA) device. The FMSA mitigates the stresses experienced by CTCs during their isolation from blood and enables viable capture. The geometric design and filtration pressures have been optimized to maximize capture efficiency, enrichment against leukocytes, and tumor cell viability. Peripheral blood as well as blood from the direct tumor environment (taken from the OR suctioning system) will be analyzed to compare the sensitivity of the FMSA and CellSearch device. Since the FMSA allows for isolation of live CTCs, they will be processed for further single cell characterization.
* Find characteristics of different CTC populations: We hypothesize that CTCs will be enriched for cancer stem cell markers as well as markers for poor prognosis and aggressive tumor growth. Our novel approach to screen and quantify a panel of biomarkers simultaneously with analysis of the CTC markers utilized by the CellSearch system to analyze of CTCs is unique. We view our assays as potential "liquid biopsies" that can screen for markers of prognosis, sensitivity to chemotherapy, response to therapy, as well as for proteins involved in proliferation, apoptosis, and immune response.

Furthermore, we plan to perform single cell analysis of gene mutations and gene expression. Next generation genomic sequencing of single CTCs may allow us to determine a genetic signature for colorectal CTCs and to identify novel biomarkers for CTC detection, disease monitoring, and therapeutic efficacy. Furthermore, the extent of heterogeneity among initially isolated CTCs, which can be compared to the primary tumor and CTCs growing in vitro, will be studied. Single CTC analysis has the potential to identify novel gene and signal transduction pathways that are activated in CTCs and to compare this genomic profile to that of the primary tumor and patient metastasis. Single cell genomic analysis in CTCs is highly innovative and will provide important information for disease monitoring as well as shed light on the underlying biology of CTCs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years will be included.
* Subjects with colorectal primary carcinomas metastatic to the liver and/or lungs who will undergo a synchronous resection of both primary tumor and liver metastases will also be enrolled.
* Subjects of all genders and ethnicities will be included.
* Subjects with the diagnosis of stage IV primary CRC will be included if metastases are limited to liver and/or lungs at the time of primary surgery.
* The histopathology of the CRC primary tumor must be documented to be adenocarcinoma.
* Subjects with the diagnosis of syn- and metachronous liver and/or lung metastases from colorectal carcinoma will be included, as long as metastases at both sites are resectable by minimal invasive or conventional approach (usually sequentially and not simultaneously).
* Liver and lung metastases must be defined according to radiological criteria. In case of doubt on radiologic findings, percutaneous biopsy will have to be obtained.
* Subjects must be capable of giving informed consent or have an acceptable surrogate capable of giving legally authorized consent on the subject's behalf.

Exclusion Criteria:

* Subjects with the concurrent diagnosis of an active second malignancy besides basal cell carcinoma of the skin will be excluded, if there is evidence of disease burden or the patient is currently treated with chemotherapy.
* Subjects with a Hemoglobin of <8g/dl in the morning of the procedure will be excluded.
* In subjects who had needed intraoperative transfusions >4 units of RPBCs, no further blood will be drawn for CTC analysis.
* Pregnant women will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with colorectal cancer metastatic to liver and/or lungs will be enrolled. Patients must be older than 18 years. No healthy volunteers/control group will be included.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Quantity of CTCs isolated during liver and/or lung metastasectomy | 1 year
  Define in which quantity CTCs are retrievable from different blood compartments and lost blood during CRC liver and lung metastases surgery using the Veridex CellSearch system and FMSA filter device

SECONDARY OUTCOMES:
Overall survival | 3 years
  Determine relationship of CTC numbers overall survival after CRC liver and lung metastases surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jussuf T Kaifi, MD PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- MS Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Result] Kaifi JT, Kunkel M, Das A, Harouaka RA, Dicker DT, Li G, Zhu J, Clawson GA, Yang Z, Reed MF, Gusani NJ, Kimchi ET, Staveley-O'Carroll KF, Zheng SY, El-Deiry WS. Circulating tumor cell isolation during resection of colorectal cancer lung and liver metastases: a prospective trial with different detection techniques. Cancer Biol Ther. 2015;16(5):699-708. doi: 10.1080/15384047.2015.1030556. PMID 25807199
- See also: PubMed link to study results — http://www.ncbi.nlm.nih.gov/pubmed/25807199
- Available data/document: Publication — http://www.ncbi.nlm.nih.gov/pubmed/25807199